CLINICAL TRIAL: NCT01178346
Title: Health-Related Quality-of-Life and Health-Care Resource Utilization Assessment in Nabi-4514 and Nabi-4515 Phase 3 Studies
Brief Title: Pharmacoeconomic Assessment in Nabi-4514 and Nabi-4515 Phase 3 Studies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: Nabi-4519
Record Dates: First submitted 2010-08-05; First posted 2010-08-10 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Smoking Cessation
Keywords: Pharmacoeconomic; Quality of Life; Health Outcomes; Smoking; NicVAX; Smoking vaccine; Smoking cessation
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NicVAX (Experimental): Experimental vaccine
  Interventions: Biological: NicVAX vaccine
- Placebo (Placebo Comparator): Placebo vaccine
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NicVAX vaccine — NicVAX vaccine given 6 times over 6 months
  Arms: NicVAX
Biological: Placebo — Placebo vaccine given 6 times over 6 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to look at pharmacoeconomic data for subjects that have received either NicVAX or placebo in the Nabi-4514 or Nabi-4515 studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are eligible for randomization or have not reached Week 12 in Nabi-4514 or Nabi-4515 studies.
* Subjects who agree to participate in health-related quality of life study.

Exclusion Criteria:

* Subjects who are unable to complete a HRQoL questionnaire because of inability to understand the language or due to mental impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of NicVAX vs. placebo on HRQoL over the study period. | one year
  QoL and health utilization questionnaires will be used to measure this outcome.

SECONDARY OUTCOMES:
To estimate utility scores for use in further health-economic models. | one year
  Scores will be computed from QoL questionnaires to measure this outcome.
To evaluate health care resource utilization. | one year
  Health care visits, medications, hospitalizations and medical procedures will be collected to measure this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Nabi Biopharmaceuticals
Locations (24):
- United States (24):
  - NicVAX Investigator, Tucson, Arizona
  - NicVAX Investigator, Encino, California
  - NicVAX Investigator, Los Alamitos, California
  - NicVAX, Newport Beach, California
  - NicVAX Investigator, San Diego, California
  - NicVAX Investigator, Denver, Colorado
  - NicVAX Investigator, Brooksville, Florida
  - NicVAX Investigator, Orlando, Florida
  - NicVAX Investigator, St. Petersburg, Florida
  - NicVAX Investigator, Tampa, Florida
  - NicVAX Investigator, Boise, Idaho
  - NicVAX, Indianapolis, Indiana
  - NicVAX Investigator, Metarie, Louisiana
  - NicVAX Investigator, Baltimore, Maryland
  - NicVAX Investigator, Minneapolis, Minnesota
  - NicVAX Investigator, Rochester, Minnesota
  - NicVAX Investigator, Omaha, Nebraska
  - NicVAX Investigator, Buffalo, New York
  - NicVAX Investigator, Cincinnati, Ohio
  - NicVAX Investigator, Mt. Pleasant, South Carolina
  - NicVAX Investigator, Nashville, Tennessee
  - NicVAX Investigator, Salt Lake City, Utah
  - NicVAX Investigator, Seattle, Washington
  - NicVAX Investigator, Madison, Wisconsin